CLINICAL TRIAL: NCT01641536
Title: An Open-label, Dose-escalating Clinical Study to Evaluate the Tolerability, Immunogenicity and Efficacy of HB-110 Administered by Electroporation (EP) in an Add-on Therapy With Entecavir in Chronic Hepatitis B Patients
Brief Title: Tolerability, Immunogenicity and Efficacy of HB-110 Administered by Electroporation in Chronic Hepatitis B Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genexine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HB110_HB_I_EP
Record Dates: First submitted 2012-06-28; First posted 2012-07-16 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Hepatitis B, Chronic
Keywords: Hepatitis, Chronic; Virus Diseases; DNA Virus Infections; Hepatitis B; Liver; Chronic Disease; HBV
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis, Chronic; Virus Diseases; DNA Virus Infections; Hepatitis B; Chronic Disease | interventions — entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1mg of HB-110 (Experimental): The subjects in this group will be administered 1 mg of HB-110 according to the protocol.
  Interventions: Genetic: HB-110
- 2mg of HB-110 (Experimental): The subjects in this group will be administered 2 mg of HB-110 according to the protocol.
  Interventions: Genetic: HB-110
- 4mg of HB-110 (Experimental): The subjects in this group will be administered 4 mg of HB-110 according to the protocol.
  Interventions: Genetic: HB-110

INTERVENTIONS:
Genetic: HB-110 — Each patient will be administered HB-110 by Electroporation for 20 weeks based on the protocol and take one pill of Entecavir(0.5 mg) per day during the study period. The Dose of HB-110 will be determined by the classical 3+3 dose escalation schedule and dose levels are 1mg, 2mg, 4mg respectively. The number of patients will be ranged from 9 to 18.
  Other Names: Baraclude(Entecavir); TriGrid™ Delivery System

SUMMARY:
This study is an open label, dose escalation study using the classical 3+3 design to determine the MTD of HB-110 and assess the safety, immunogenicity and efficacy of HB-110 DNA therapeutic vaccine administered by Electroporation in combination with Entecavir in chronic hepatitis B patients.

DETAILED DESCRIPTION:
The patients enrolled in the trial will be successively allocated into three cohorts for HB-110 1mg, 2mg, and 4mg in combination with Entecavir according to the classical 3+3 protocol design. They will be administered by Electroporation device.

The scheduled assessments and visits will be carried out over three periods: run-in period, treatment period, and follow-up period.

The run-in period includes the screening visit where a written informed consent is obtained and the screening period where patients are assessed for eligibility. It will be completed within 14 days prior to Visit 1. The patients meeting inclusion criteria will start the treatment period.

During the treatment period, subjects will be administered HB-110 by Electroporation at each visit in combination with antiviral drug, Entecavir.

The Follow-up period starts once subjects complete the treatment period and will continue until the follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Agreed that female subjects or female partners of male subjects will not be pregnant during the study.
* Chronic hepatitis B patients who are taking Entecavir at the Screening Visit for 6 months or longer
* Have not used IFN alpha or antiviral drugs within the previous 6 months for treating hepatitis.
* Have blood HBV DNA level of ≤300 copies/mL determined at Screening Visit
* Have an ALT level less than or equal to 2 times the upper limit of normal [ULN] at the Screening Visit
* Provide a signed voluntary written informed consent for study participation

Exclusion Criteria:

* Who have participated in other studies within previous 30 days from Screening Visit
* Have the following decompensated liver parameters,

  * serum albumin level <3 g/dL,
  * total bilirubin level >2.5 mg/dL,
  * international normalized ratio (INR) >1.8
* Do not have adequate renal function as determined by serum creatinine level 1.5 times more than normal range(1.2 mg/dL)
* Had a previous liver transplant or bone marrow transplant
* Are currently taking immunosuppressive or possible immunomodulatory drugs
* Women who are pregnant or breastfeeding
* female subjects will be pregnant or breastfeed during the study
* History of allergy/hypersensitivity to drugs
* Any clinically significant acute or chronic unstable renal, cardiac or endocrine disease (e.g., cardiac failure, renal failure, pancreatitis, diabetes mellitus)
* Presence of any other primary or secondary hepatic disease (e.g., hemochromatosis, Wilson's disease, alcoholic hepatic disease, non alcoholic fatty liver, alpha-1-antitrypsin deficiency and so on) other than hepatitis B
* Who were observed for hepatocellular mass by ultrasonography and have an abnormal increase of serum AFP
* Past or present history of hepatocarcinoma
* History of grand mal epilepsy, or currently on anti-epileptic medications
* Occurrence of at least one episode of syncope within the last 12 months
* Presence of an implantable cardiac device (pacemaker, automated implantable cardioverter defibrillator [AICD]) or implantable nerve stimulator
* Who have arrhythmia
* Any other conditions that are considered inappropriate for the study by the Investigator.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Frequency of Adverse Events | 1 year
Degree of Adverse Events | 1 year

SECONDARY OUTCOMES:
Level of HBV antigen-specific T-cell ex-vivo ELISPOT | 1 year
Level of HBV antigen-specific T-cell cultured ELISPOT | 1 year
Maintenance of HBeAg seroconversion if they had HBeAg seroconversion at Screening Visit, otherwise occurence of HBeAg seroconversion at Follow-up Visit | 1 year
HBsAg loss and HBsAg seroconversion rate at Follow-up Visit | 1 year
ALT level | 1 year
level of HBsAg titer | 1 year
Number of HBV DNA Copies | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Kew Yoon, M.D., Principal Investigator — The Department of Gastroenterology at Seoul St. Mary's Hospital
Locations (1):
- Seoul St. Mary's Hospital, Seoul, South Korea